CLINICAL TRIAL: NCT03499769
Title: Comparison of NOSE and Conventional Methods in Laparoscopic Total Colon Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Ersin Gündoğan, operator doctor, Inonu University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2018/3-3
Record Dates: First submitted 2018-03-27; First posted 2018-04-17 (Actual); Last update posted 2018-07-20 (Actual); Status verified 2018-02

CONDITIONS: Surgical Incision
MeSH Terms: conditions — Surgical Wound | interventions — Natural Orifice Endoscopic Surgery; Congresses as Topic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- natural orifice (Experimental): Patients who underwent laparoscopic surgery and removed the specimen from the natural orifice will be gathered. demographic data and perioperative results will be compiled
  Interventions: Procedure: natural orifice
- conventional (No Intervention): patients who underwent laparoscopic surgery and removed specimen with conventional will be gathered. demographic data and perioperative results will be compiled. (conventional extraction is suprapubic or median incision)

INTERVENTIONS:
Procedure: natural orifice — laparoscopic total colon surgery and patients who are removed from the natural orifice and conventional will gather
  Other Names: conventional
  Arms: natural orifice

SUMMARY:
Laparoscopic total colectomy (LTC) is an accepted surgical procedure for several colonic pathologies. Additionally, specimen extraction through the natural orifices is an emerging method when combined with the totally laparoscopic procedures. Our observations on natural orifice surgery was promising . In our daily surgical practice, investigators prefer the intracorporeal anastomosis and this study was conducted to compare the specimen extraction sites after LTC. Here investigators aimed to compare the results of conventional and natural orifice specimen extractions (NOSE) after totally LTCs.

DETAILED DESCRIPTION:
compare the patient-selected NOSE method and conventional method in laparoscopic total colon surgery

ELIGIBILITY:
Inclusion Criteria:

* laparoscopic total colectomy patients

Exclusion Criteria:

* no

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2017-12-25 (Actual); Study Completion 2017-12-28 (Actual)

PRIMARY OUTCOMES:
Visual Analog Score | 240 days
  Visual Analog Score for pain (1-10 score)

CONTACTS AND LOCATIONS:
Overall Officials: Ersin Gündoğan, Principal Investigator — Inonu Unıversity- general surgery
Locations (1):
- Inonu University, Malatya, Turkey (Türkiye)